CLINICAL TRIAL: NCT00150696
Title: Risedronate for Prevention of Osteoporosis After Spinal Cord Injury
Brief Title: Risedronate for the Prevention of Osteoporosis in People With Spinal Cord Injury.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); St. Joseph's Healthcare Foundation (Other); Queen Elizabeth Hospital NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TRI REB #02-040; ONRO-79
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Acute Spinal Cord Injury.
Keywords: Osteoporosis; Spinal Cord Injury
MeSH Terms: conditions — Osteoporosis; Spinal Cord Injuries | interventions — Risedronic Acid

INTERVENTIONS:
Drug: Risedronate

SUMMARY:
The purpose of this study is to find out if Risedronate works to prevent osteoporosis after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury less than 100 days.
* Must be able to swallow tablets and sit upright.

Exclusion Criteria:

* Bilateral knee flexion contractures.
* Pregnant, lactating or post-menopausal females.
* Paget's disease, osteomalacia, steroid induced bone loss, untreated thyroid disease, iritis, uveitis, pancreatitis, gastritis, peptic ulcer or cholecystitis.
* Treatment in the last year with calcitonin, fluoride or anabolic steroid.
* Concurrent treatment with prednisone.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38
Dates: Start 2000-02; Study Completion 2005-11

PRIMARY OUTCOMES:
Change in bone mineral density of the distal femur and proximal tibia between baseline, 12-months and 24-months.

SECONDARY OUTCOMES:
Change in bone mineral density of the total body, spine and femoral neck between baseline, 12-months and 24-months.
Change in biochemical markers of bone turnover between baseline, 12-months and 24-months.
Frequency and severity of adverse events.
Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: B. Cathy Craven, MD, FRCPC, Principal Investigator — Toronto Rehabilitation Institute
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Chedoke Site, Hamilton, Ontario
  - Toronto Rehab, Lyndhurst Centre, Toronto, Ontario